CLINICAL TRIAL: NCT02736630
Title: National Epidemiology Survey on the Incidence of Perioperative Hypothermia in Patients With Elective Surgery Under General Anesthesia in Turkey
Brief Title: Incidence of Perioperative Hypothermia in Patients With Elective Surgery Under General Anesthesia in Turkey
Acronym: GAPOHI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Collaborators: Uludag University (Other)
Responsible Party: Principal Investigator, Hulya Bilgin, Prof, Turkish Society of Anesthesiology and Reanimation
Other Study IDs: TurkishARD
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Perioperative Hypothermia
Keywords: general anaesthesia; elective surgery; national epidemiology; turkey
MeSH Terms: interventions — Body Temperature

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: body temperature — intermittant tympanic temperature measurement during surgery

SUMMARY:
Primary objective of the study is to project the incidence rate of perioperative hypothermia under general anesthesia in patients who go under minimum 1 hour long elective surgery in at least 25 hospitals/medical centers in Turkey .

Secondary objectives are to determine the patient risk factors associated with perioperative hypothermia, to determine the surgery risk factors associated with perioperative hypothermia, to determine the other risk factors associated with perioperative hypothermia, intraoperative infusion volume and effect of warming, intraoperative irrigation volume and effect of warming, intraoperative blood infusion volume and effect of warming, to determine complications related to perioperative hypothermia, to improve patient temperature management awareness and processes.

DETAILED DESCRIPTION:
Mild hypothermia during perioperative period is very common, and the percentage accounts for about half of all patients undergoing operations, which is directly related to the following three major adverse events that significantly increase their risks: 1) cardiac complications, 2) hemorrhage, 3) infection complications , particularly in patients with high risk factors (ASA grade III, IV). Furthermore, the decrease in body temperature may also lead to the following situations: 1) prolongation in retention time in post-anesthetic ICU (PACU), 2) decrease in the thermal comfort for patients, and thus affecting the satisfaction degree of patients and increasing cost.

From the viewpoint of patient safety, body surface temperature is only a vital sign. Therefore, in order to prevent hypothermia during perioperative period, core temperature monitoring must be carried out from the very beginning of the operation. The heat loss during operations should be minimized. Active warming measurements should be taken for high risk patients during the entire procedures of operations.

Although the literature have reported high incidence rate of hypothermia during perioperative period of selective operations, there's no detailed information about perioperative hypothermia prevalence in Turkey. Actually there are only a few studies about patient warming effectiveness. A small scale study done by Kocaeli University in Turkey in 2013 shows the post operative hypothermia incidence as 45.7%. Another study and survey done by Cerrahpasa Medicine Faculty shows even among healthcare professionals there is great variance about the perception and results of hypothermia. Those facts drives investigators to gather more clinical evidence about perioperative hypothermia.

Under the supervision of Turkish Anesthesiology and Reanimation Society and coordination of Prof Dr Hulya Bilgin from Uludag University Medicine Faculty Anesthesiology and Reanimation Clinic it is aimed to gather evidence about hypothermia prevalence patients who go under minimum 1 hour elective surgery under general anesthesia. So with the results of such a study it is aimed to improve the standard protocols regarding patient temperature management, patient warming management and also to avoid the complications and costs related to hypothermia.

In order to further obtain information on the current status of temperature monitoring and perioperative warming practice in most parts of the country, to project incidence rate of perioperative hypothermia in most parts of the country, explore the relationship between perioperative hypothermia and postoperative clinical outcome, and to provide evidence for the improvement of perioperative body temperature management guidelines in accordance with characteristics of the current Turkish healthcare status, investigators will conduct surveys in department of anesthesiology over certain regions of Turkey to carry out a large scale prospective study. In the study, investigators will search the incidence rate of perioperative hypothermia in the surveyed areas, explore the causes of hypothermia, base on which it is expected to enable to project perioperative hypothermia incidence rate, to verify the effectiveness of perioperative hypothermia risk assessment questionnaire for patients under general anesthesia, and to provide guidance and evidence for the clinical practice of perioperative warming care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years old
* Subject will undergo an elective surgery under general anesthesia
* The duration of surgery is expected to be over 60 minutes
* Patients or relatives whom the study is explained and their informed consent is documented
* Patients who are preplanned to be in ICU after surgery will not be excluded

Exclusion Criteria:

* Central high fever caused by enter nerves system disease or condition, including that induced by cerebrovascular disease, cerebral trauma, cerebral surgeries, epilepsy and acute hydrocephalus
* Thermoregulation abnormalities including malignant hyperthermia (MHS) and neuroleptic malignant syndrome, hypothyroidism or hyperthyroidism diagnosed by substantial evidence
* Infectious fever
* Temperature is higher than 37.8 Celcius degree within 3 days before surgery
* Diseases or that may lead to inaccuracy in measurement, such as ear infection
* Therapeutic preoperative hypothermia
* Trauma related bleeding, shock and extensive fluid resuscitating surgeries
* Acute or chronic spine injury cases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of perioperative hypothermia in Turkey | 2 months

SECONDARY OUTCOMES:
The patient risk factors associated with perioperative hypothermia. | 2 months
The surgery risk factors associated with perioperative hypothermia. | 2 months
Complications related to perioperative hypothermia | 2 months
Patient temperature management development strategies | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Bilgin, Prof, Principal Investigator — Turkish Society of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Smith JJ, Bland SA, Mullett S. Temperature--the forgotten vital sign. Accid Emerg Nurs. 2005 Oct;13(4):247-50. doi: 10.1016/j.aaen.2005.08.002. Epub 2005 Sep 30. PMID 16199165
- [Background] Sessler DI. Complications and treatment of mild hypothermia. Anesthesiology. 2001 Aug;95(2):531-43. doi: 10.1097/00000542-200108000-00040. No abstract available. PMID 11506130
- [Result] Doufas AG. Consequences of inadvertent perioperative hypothermia. Best Pract Res Clin Anaesthesiol. 2003 Dec;17(4):535-49. doi: 10.1016/s1521-6896(03)00052-1. PMID 14661656
- [Result] Mahoney CB, Odom J. Maintaining intraoperative normothermia: a meta-analysis of outcomes with costs. AANA J. 1999 Apr;67(2):155-63. PMID 10488289